CLINICAL TRIAL: NCT07000916
Title: Medical Follow-up of New Cases of Polyarthritis in Children and Young Adults. Optimization of Clinical Response, Remission, Quality of Life and Analysis of Prognostic Markers
Brief Title: Medical Follow-up of New Cases of Polyarthritis in Children and Young Adults
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Cap 48 polyarthrite
Record Dates: First submitted 2019-04-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Juvenile Idiopathic Arthritis; Rheumatoid Arthritis; Psoriatic Arthritis; Systemic Lupus Erythematosus; Diffuse Systemic Sclerosis; Seronegative Arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis, Rheumatoid; Arthritis, Psoriatic; Lupus Erythematosus, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — residual blood and urine sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- juvenile idiopathic arthritis (JIA): aged <= 16 y.o. recent diagnosis of JIA and DMARDs treatment-naive patients; aged <18 y.o. recent diagnosis of JIA
- rheumatoid arthritis (RA): aged =>18; =< 50 y.o. recent diagnosis of RA and DMARDs treatment-naive patients
- diffuse systemic sclerosis (dSS): aged =>18; =< 50 y.o. recent diagnosis of dSS and DMARDs treatment-naive patients
- seronegative arthritis (UA): aged =>18; =< 50 y.o. recent diagnosis of UA and DMARDs treatment-naive patients
- systemic lupus erythematosus (SLE): aged =>18; =< 50 y.o. recent diagnosis of SLE and DMARDs treatment-naive patients

SUMMARY:
Population:

Juvenile idiopathic arthritis (JIA), rheumatoid arthritis (RA) and seronegative / psoriatic / undifferentiated arthritis (UA), systemic lupus erythematosus (SLE) or diffuse systemic sclerosis dSS).

Naïve to basic treatment OR treated for ≤ 3 months; except for patients with JIA.

These 5 cohorts will be subject to standardized clinical monitoring.

DETAILED DESCRIPTION:
This study is proposed by the Rheumatology and Pediatrics departments of the 3 French-speaking Universities.

The first objective will be to include a progressive number of new young patients (≤ 50 years) in order to optimize and standardize care and clinical response objectives. The number of 25% of new incident cases will be sought with an increase of 20% each year during the 5 to 10 years of this project.

Population: JIA, RA/UA, SLE, dSS (American Congres of Rheumatology criteria). Naïve to basic treatment OR treated for ≤ 3 months; except for patients with JIA.

These 5 cohorts will be subject to standardized clinical monitoring and specific objectives that will make it possible to analyze the number of patients with a good control of the disease and/or a clinical remission, defined according to the international criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of juvenile idiopathic arthritis, rheumatoid arthritis and seronegative / psoriatic / undifferentiated arthritis, systemic lupus erythematosus or diffuse systemic sclerosis (ACR criteria).
* Naïve to basic treatment OR treated for ≤ 3 months; except for patients with JIA.

Exclusion Criteria:

* Treated for > 3 months
* > 50 years old

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with juvenile idiopathic arthritis, rheumatoid arthritis and seronegative / psoriatic / undifferentiated arthritis, systemic lupus erythematosus or diffuse systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-09-11 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate or absence of synovitis in Rheumatoid arthritis patients | Through the entire study, during approximately 15 years

OTHER OUTCOMES:
Remission rates improvement in Juvenile arthritis (JIA) patients | Through the entire study, during approximately 15 years
Reduction in damage rate in Systemic Lupus Erythematosus patients | Through the entire study, during approximately 15 years
Inclusion of at least 80% of the incident cases of diffuse Systemic sclerosis | Through the entire study, during approximately 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, Pr, Study Director — UCLouvain - IREC
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No